CLINICAL TRIAL: NCT06837870
Title: A Randomized Comparison of Percutaneous Closure to a Figure-of-eight Suture With Manual Compression for Hemostasis of Large-bore Access for Leadless Pacemaker Implantation
Brief Title: Percutaneous Closure Versus Figure-of-eight Suture for Hemostasis in Leadless Pacemaker Implantation.
Acronym: PERCLOSE-LP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Soroosh Kiani, Assistant Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002172
Record Dates: First submitted 2025-01-30; First posted 2025-02-20 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Vascular Closure; Pacemaker Implantation; Leadless Pacemaker
Keywords: perclose; percutaneous closure; leadless pacemaker; venous access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SMC (Experimental): Percutaneous suture mediated closure group
  Interventions: Device: percutaneous suture mediated closure
- MC (Active Comparator): Manual Compression (with a figure-of-eight) closure group (i.e., control).
  Interventions: Device: Figure of Eight Suture

INTERVENTIONS:
Device: percutaneous suture mediated closure — Vascular closure with a commercially available SMC device.
  Other Names: PerClose, ProStyle
  Arms: SMC
Device: Figure of Eight Suture — Manual Compression with Figure of Eight Suture (control).
  Other Names: Fo8
  Arms: MC

SUMMARY:
The study will be a randomized comparison of percutaneous suture-mediated closure (SMC) versus manual compression with a superficial figure-of-eight suture (MC) for large bore venous access used for leadless pacemaker implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older
* Patients undergoing leadless pacemaker implant at UMass Chan Medical Center
* Subjects able to understand and provide written informed consent.

Exclusion Criteria:

* Patients who are pregnant
* Patents who are not able to ambulate prior to the procedure
* Other conditions that, in the opinion of the investigator constitute a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation
* Prisoners or wards of the state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Time to Hemostasis | During the procedure.
  Time from sheath pull to hemostasis.

SECONDARY OUTCOMES:
Time to discharge eligibility | Periprocedurally, from day 0 up to discharge; typically 0-1 days but up to the time of hospital discharge.
  Time from sheath pull to eligibility for discharge.
Major access related complications | 0 and 30 days
  Composite and individual access related complications
Minor access related complications | 0 and 30 days
  Composite and individual access related complications
Patient reported outcomes | 0 and 30 days
  Patient reported outcomes of both a pain and satisfaction ascertained by a questionnaire reported as a total/composite score of all questions, as well as the score for each individual question on the questionnaire (rated on a likert scale).
Costs | 0 and 30 days
  Direct and indirect procedure and peri-procedural cost data

OTHER OUTCOMES:
Time to Ambulation | Periprocedurally. Periprocedurally, from day 0 up to discharge; typically 0-1 days but up to the time of hospital discharge.
  Time from sheath pull to ambulation

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No